CLINICAL TRIAL: NCT02017262
Title: Group Self-Management for Persons With Depression and Medical Illness
Brief Title: Group Self-Management of Depression and Medical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Isabel T. Lagomasino, MD, MSHS, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH093557 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Depression; Chronic Disease; Hispanic Americans
Keywords: Self-care; Patient education
MeSH Terms: conditions — Depression; Chronic Disease | interventions — Self Care; Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-management group (Experimental): 8 weekly sessions of group self-management
  Interventions: Behavioral: Self-management group
- Enhanced usual care (Active Comparator): Usual care by primary care provider, plus educational pamphlet about depression, list of local mental health resources, and letter for provider advising him/her of depression diagnosis
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Self-management group — 8 weekly sessions of group self-management
  Other Names: Self-care; Patient education
  Arms: Self-management group
Behavioral: Enhanced usual care — Usual care by primary care provider, plus educational pamphlet about depression, list of local mental health resources, and letter for provider advising him/her of depression diagnosis
  Arms: Enhanced usual care

SUMMARY:
This project addresses the important public health need to reduce ethnic disparities in depression care by pilot testing and refining a culturally tailored, low-cost intervention for improving both depression and general medical outcomes among Latinos in safety net primary care settings. Cuerpo Sano, Mente Sana is a newly developed, lay-led, group self-management intervention that educates and empowers patients in their own health care and has the potential for widespread implementation and sustainability in primary care because it is responsive to patient, provider, and system preferences and needs. After completing an assessment of study clinic sites, we will conduct a pilot test of Cuerpo Sano, Mente Sana with 30 low-income, Spanish-speaking primary care patients. After reviewing pilot findings, we will revise the intervention and study plan, and will conduct a second pilot trial. After reviewing findings from this second trial, we will finalize the intervention and study plan in preparation for larger studies to test Cuerpo Sano, Mente Sana versus other interventions for addressing depression among Latinos in safety net primary care.

DETAILED DESCRIPTION:
Latinos suffer a greater disability burden from depression than whites due to low rates of quality depression care. Depression is common among Latinos in primary care settings and is also often chronic, recurring, and comorbid with chronic medical illness. Improving outcomes for both depression and chronic medical illness requires patients to become educated, active partners in managing their illnesses. Latinos desire education regarding general and mental health; have stigma-related concerns regarding mental health care; and prefer psychotherapy to medication. However, safety net primary care providers and clinics often prioritize improving medical outcomes and lack the resources for depression care, especially psychotherapy. There is an important public health need to develop a culturally tailored, low cost intervention that includes educational and psychotherapeutic elements, targets medical illness and depression, and destigmatizes depression care.

In response to patient, provider, and clinic preferences and resources for depression care, we developed but have not yet tested an innovative, theoretically-based group intervention, drawing upon two evidence-based interventions that improve self-efficacy: group cognitive behavioral therapy (CBT) for depression and group self-management for chronic medical illness. Professionally-led group CBT is effective for depression among ethnic minorities in primary care but is difficult to sustain. Among patients with chronic medical illness, lay-led group self-management programs educate and empower patients to engage in healthful behaviors and participate in their care. The groups improve self-efficacy, health-related behaviors, and outcomes; have been adapted for diverse conditions; and have been widely disseminated and sustained. However, standard self-management groups do not improve depression. We thus enhanced the Spanish-language Tomando Control de su Salud chronic disease self-management program by adding depression-related educational and skill-building content from group CBT.

We will pilot test and refine Cuerpo Sano, Mente Sana, our newly enhanced self-management program for depression and chronic medical illness. Following a framework for successful implementation of interventions, we will 1) evaluate intervention context and refine our intervention and implementation strategy; 2) conduct a randomized trial with 30 low-income Spanish-speaking patients with depressive disorder and chronic medical illness; 3) review pilot findings of feasibility, implementation, and potential sustainability with a multistakeholder panel and then revise our materials and procedures; 4) conduct a second trial with 30 additional patients; and 5) review additional pilot findings (including 3- and 6-month intervention effects on self-efficacy, self-care behaviors, and depression and health outcomes and interviews with clinic stakeholders) and finalize the intervention and implementation strategy. This study lays the groundwork for future comparative effectiveness studies of strategies to address depression among Latinos in safety net primary care.

ELIGIBILITY:
Inclusion Criteria:

* Established primary care patient
* Spanish-speaking
* Depression (major depression, dysthymia, minor depression)
* Chronic medical illness (diabetes, hypertension, dyslipidemia, heart disease, lung disease, cerebrovascular disease, arthritis)

Exclusion Criteria:

* Bipolar disorder
* Psychosis
* Cognitive impairment
* Active suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Depressive symptom severity (Hopkins Symptoms Checklist, or SCL) | Change from baseline in depressive symptom severity at 3-months

SECONDARY OUTCOMES:
Health-related quality of life (Short-Form-12) | Change from baseline in health-related quality of life at 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Megan Dwight-Johnson, MD MPH, Principal Investigator — VA Medical Center-West Los Angeles
Locations (1):
- LAC+USC Medical Center, Primary Care Clinics, Los Angeles, California, United States